CLINICAL TRIAL: NCT06033040
Title: Clinical Study on the Diagnostic and Predictive Value of MRI Multifunctional Imaging in Bladder Tumors
Brief Title: Medical Imaging in Bladder Tumors by MRI
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Sponsor
Other Study IDs: SYSKY-2023-549-01
Record Dates: First submitted 2023-07-27; First posted 2023-09-13 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Bladder Tumor; Magnetic Resonance Imaging
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: MRI — Functional sequence imaging (MDME, IVIM) sequences were added to the routine MRI scan of patients with bladder tumor

SUMMARY:
This study prospectively included 178 patients with bladder neoplastic lesions who planned to undergo surgery (with or without preoperative neoadjuvant chemotherapy). Inclusion criteria: Patients with pathologically confirmed bladder cancer after radical or partial cystectomy or TURBT (< 2 weeks between surgical resection and imaging). Exclusion criteria: 1) Prior history of chemotherapy and/or radiotherapy; 2) No surgical resection; 3) The interval between surgical resection and imaging examination is > 2 weeks; 4) Obvious artifacts; 5)MRI scan contraindications. All subjects underwent pelvic MRI. Data was collected using a Siemens VIDA 3TMR scanner (Siemens Healthcare, Erlangen, Germany). All subjects underwent standardized scanning protocols. The obtained images are post-processed and the experimental results are analyzed statistically.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical diagnosis of bladder neoplasm
2. Must undergo radical or partial cystectomy or TURBT surgery within 2 weeks between surgical resection and imaging

Exclusion Criteria:

1. A history of pelvic radiotherapy or chemotherapy;
2. Lack of pathological findings or no surgery;
3. The interval between surgical resection and imaging examination > 2 weeks;
4. Poor image quality due to poor coordination or motion artifacts;
5. MRI scan contraindications

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Patients with bladder neoplasm planned to undergo surgery
Sampling Method: Probability Sample
Enrollment: 178 (Estimated)
Dates: Start 2023-08-15 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
quantitative parameters by MRI | From the time the participants completed the MRI scan to the post-processing of the resulting images,assessed up to 2 months
  quantitative parameters by functional MRI

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen Memorial Hospital, Sun Yat-sen University, Guangzhou, Guangdong, China